CLINICAL TRIAL: NCT03443778
Title: Comparison of Peritonsillar Dexamethasone-bupivacaine and Bupivacaine Infiltration for Tonsillectomy Pain Relief in Children:a Randomized,Double Blind,Controlled Study.
Brief Title: Dexamethasone-bupivacaine Versus Bupivacaine for Tonsillectomy Pain.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Leyla Kılınc, Principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 907-12.12.2017
Record Dates: First submitted 2017-12-27; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Tonsillectomy
Keywords: tonsillectomy pain; dexamethasone; bupivacaine
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nacl 0,9% (Control) group (Active Comparator): Nacl 0,9% 3-5 ml separately two part for each tonsil before surgery
  Interventions: Drug: Nacl 0,9 %
- Bupivacaine 0,5% (Active Comparator): Bupivacaine 0.5% 1 mg/kg with in Nacl 0,9% 3-5 ml separately two part for each tonsil before surgery
  Interventions: Drug: Bupivacaine 0.5%
- Bupivacaine 0,5% , Dexamethasone (Active Comparator): Bupivacaine 0,5% 1 mg/kg,dexamethasone 0.5 mg/kg (max dosage 8mg) 3-5 ml separately two part for each tonsil before surgery
  Interventions: Drug: Bupivacaine 0.5% , Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine 0.5% — Marcaine 0.5% Injectable Solution
  Other Names: Marcaine 0,5%
  Arms: Bupivacaine 0,5%
Drug: Bupivacaine 0.5% , Dexamethasone — Bupivacaine 0.5% , Dexamethasone
  Other Names: Dekort; Marcaine 0,5 % Injectable Solution
  Arms: Bupivacaine 0,5% , Dexamethasone
Drug: Nacl 0,9 % — Injectable Solution
  Other Names: Serum Physiologic
  Arms: Nacl 0,9% (Control) group

SUMMARY:
Investigators compared in this study peritonsillar infiltration of bupivacaine %0.5 (n=40 participants) versus bupivacaine % 0.5 and dexamethasone (number 40participants ) before surgery for reduce posttonsillectomy pain.And control group (n= 40participants) participants received peritonsillar Nacl 0,9% .

DETAILED DESCRIPTION:
Bupivacaine hydrochloride amid structure,long acting local anesthetic. Dexamethasone has strong anti-inflammatory drug reduce postoperative pain and nause and vomiting.Preoperative iv dexamethasone is routinely using for reduce tonsillectomy pain.Lots of studies show that adding dexamethasone to local anesthetic at peripheral nerve block prolongs the analgesic effect.Also preoperative iv dexamethasone prolongs the analgesic effects of local anesthetic infiltration .

Post tonsillectomy pain still a serious problem ,it effects postoperative morbidity.Different medicine combination used to applies for peritonsillar infiltration and multimodal iv and oral medication to reduce posttonsillectomy pain.İn this study investigators will use iv dexamethasone for all participants and investigators hypothesis that adding dexamethasone to bupivacaine for peritonsillar infiltration will reduce postoperative pain scores , consumption of rescue analgesic ,patient and family satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Tonsillectomy surgery for recurrent tonsillitis Sleep disorder breathing

ExclusionCriteria:

Patients with active upper respiratory tract infection Patients with significant cognitive impairment Bupivacaine hypersensitivity Dexamethasone hypersensitivity Taking chronic systemic steroids

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-03-15 (Estimated); Study Completion 2018-04-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of moderate/severe pain(>/= 4 of 10 Pain Scores) | postoperative 7day .
  Pain Scores will measure ; Face, Leg, Activity, Cry, Consolability score (FLACC) Interpreting the Score 0 Relaxed & comfortable
  1 - 3 = Mild discomfort 4 - 6 = Moderate pain 7 -10 = Severe pain or discomfort or both . 0 score is the best ,10 score is the worse score. 4 and up scores will considered to be the range to be treated .Pain score will measure at home ; Face Pain Scale 0 no pain 10 worse pain. Every day in the morning after phone call pain scores will ask patient/patient guardians. 4 and up scores will treated

SECONDARY OUTCOMES:
Side effects (nause,vomiting) | postop seven day
  Nause will measure with visual analog scale (VAS) . 0 is the best 10 is the worse score. vomiting will measure with present/absent
Rescue analgesic consumption at PACU (post-anaesthesia care unit) | At Pacu 1 hour
  Pain Scores will measure ; Face, Leg, Activity, Cry, Consolability score (FLACC) Interpreting the Score 0 Relaxed & comfortable
  1 - 3 = Mild discomfort 4 - 6 = Moderate pain 7 -10 = Severe pain or discomfort or both . 0 score is the best ,10 score is the worse score. 4 and up scores will considered to be the range to be treated with iv paracetamol (10 mg/kg maximum Daily dosage) . İf the pain score is still 4 and up it will treated with tramadol 1 mg/kg).
Rescue analgesic consumption first day at hospital | 4,8,12,24 h at hospital in first postoperative day.
  Pain Scores will measure ; Face, Leg, Activity, Cry, Consolability score (FLACC) Interpreting the Score 0 Relaxed & comfortable
  1 - 3 = Mild discomfort 4 - 6 = Moderate pain 7 -10 = Severe pain or discomfort or both . 0 score is the best ,10 score is the worse score. 4 and up scores will treated with oral paracetamol (10 mg/kg)
Rescue analgesic consumption at home | postop 2-3-5-6- 7. day
  Pain Scores will measure ; Face Pain Scale 0 no pain 10 worse pain. 4 and up scores will treated with oral paracetamol (10 mg/kg)
Parents satisfaction | postop seven day
  Parents satisfaction will measure visual analog scale (VAS) . 0 is the best 10 is the worse score.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Kilinc, Md, Study Director — Md
Locations (1):
- Leyla Kilinc, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant (IPD) to the other researchers

REFERENCES:
- [Background] Bayram A, Dogan M, Cihan C, Karatas D, Gokahmetoglu G, Ozcan I. The Efficacy of Levobupivacaine Hydrochloride-Dexamethasone Infiltration for Post-Tonsillectomy Pain in Adults. J Craniofac Surg. 2015 Oct;26(7):e651-3. doi: 10.1097/SCS.0000000000001975. PMID 26468853
- [Background] Basuni AS, Ezz HA, Albirmawy OA. Preoperative peritonsillar infiltration of dexamethasone and levobupivacaine reduces pediatric post-tonsillectomy pain: a double-blind prospective randomized clinical trial. J Anesth. 2013 Dec;27(6):844-9. doi: 10.1007/s00540-013-1638-0. Epub 2013 May 25. PMID 23708881